CLINICAL TRIAL: NCT02078986
Title: Comparison of the Effect of Whole-Body Electromyostimulation Versus High Intensity Resistance Exercise Training on Body Composition and Strength in Middle Aged Males
Brief Title: Effectiveness of WB-EMS Versus HIT-Resistance Training (RT)
Acronym: EMSvsHIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Klinikum Nürnberg (Other); Benevital Health Park, Herzogenaurach (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Professor Dr. Wolfgang Kemmler, PhD, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMSvsHIT; IMP_FAU (Other: Institute of Medical Physics, University of Erlangen-Nuremberg)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Healthy; Sedentary; Untrained
Keywords: Whole-Body-Electromyostimulation; High Intensity Resistance Exercise Training (HIT); Lean Body Mass; Muscle Strength
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Body Electromyostimulation (Experimental)
  Interventions: Other: Whole Body Electromyostimulation
- High Intensity Resistance Exercise Training (Experimental): Supervised High Intensity Resistance Exercise 2-3 session/week/14 weeks
  Interventions: Other: High Intensity Resistance Exercise Training

INTERVENTIONS:
Other: Whole Body Electromyostimulation — Supervised WB-EMS, 3 sessions in 2 weeks (1,5 sessions/week) for 14 weeks
  Arms: Whole Body Electromyostimulation
Other: High Intensity Resistance Exercise Training — Supervised High Intensity Resistance Exercise Training (HIT) 2-3 sessions/week for 14 weeks
  Arms: High Intensity Resistance Exercise Training

SUMMARY:
The main aim of the study is to determine the effects of Whole-Body Electromyostimulation (WB-EMS) on body composition and muscle strength compared with the "golden standard" High Intensity Resistance Exercise Training (HIT) in healthy sedentary middle aged males.

ELIGIBILITY:
Inclusion Criteria:

* male, 25 to 55 years old
* sedentary / untrained
* Body Mass Index 20 - 30 kg/m2

Exclusion Criteria:

* absent ≥ 2 weeks during the interventional period
* medication or diseases with relevant impact on muscle metabolism
* conditions that prevent WB-EMS (e.g. epilepsy, cardiac pacemaker)
* severe neurological diseases

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Lean Body mass | 14 weeks (baseline to 14 week follow-up assessment)
  Lean Body Mass as assessed by Dual Energy x-Ray Absorptiometry (DXA) was determined twice, at baseline and after 14 weeks of exercise (WB-EMS or HIT)

SECONDARY OUTCOMES:
Appendicular Skeletal Muscle Mass | 14 weeks (baseline to 14 week follow-up assessment)
  Appendicular Skeletal Muscle Mass (ASMM) as assessed by DXA was determined at baseline and after 14 weeks of exercise (WB-EMS or HIT)

OTHER OUTCOMES:
Isokinetic Muscle Strength of the leg extensors and -flexors | 14 weeks (baseline to 14 week follow-up assessment)
  Isokinetic Muscle Strength leg extensors and -flexors as assessed by a an isokinetic leg press was determined at baseline and after 14 weeks of exercise (WB-EMS or HIT).

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang K Kemmler, PhD, Study Chair — Institute of Medical Physics, University of Erlangen-Nuremberg; Simon O von Stengel, PhD, Study Director — Institute of Medical, University of Erlangen-Nuremberg; Marc Teschler, MA, Principal Investigator — Institute of Medical Physical, University of Erlangen-Nuremberg
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nuremberg, Erlangen, Franconia, Germany

REFERENCES:
- [Background] Kemmler W, von Stengel S. Whole-body electromyostimulation as a means to impact muscle mass and abdominal body fat in lean, sedentary, older female adults: subanalysis of the TEST-III trial. Clin Interv Aging. 2013;8:1353-64. doi: 10.2147/CIA.S52337. Epub 2013 Oct 7. PMID 24130433
- [Background] Kemmler W, von Stengel S. Alternative Exercise Technologies to Fight against Sarcopenia at Old Age: A Series of Studies and Review. J Aging Res. 2012;2012:109013. doi: 10.1155/2012/109013. Epub 2012 Feb 20. PMID 22500224
- [Background] Kemmler W, Bebenek M, Engelke K, von Stengel S. Impact of whole-body electromyostimulation on body composition in elderly women at risk for sarcopenia: the Training and ElectroStimulation Trial (TEST-III). Age (Dordr). 2014 Feb;36(1):395-406. doi: 10.1007/s11357-013-9575-2. Epub 2013 Aug 16. PMID 23949160
- See also: Related Info — http://www.imp.uni-erlangen.de/